CLINICAL TRIAL: NCT04147572
Title: Inspiratory Flow Parameters With Placebo Tiotropium Easyhaler® and Placebo Spiriva® Capsule Via HandiHaler® in Patients With COPD and in Healthy Volunteers. Substudy: Easyhaler® and HandiHaler® Usability Study in Patients With COPD
Brief Title: Inspiratory Flow Parameters With Placebo Easyhaler and Placebo HandiHaler
Acronym: TIOPIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3122004
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteer; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Inhaler A, Tiotropium Easyhaler (Experimental): Placebo Tiotropium Easyhaler, type A
  Interventions: Drug: Placebo Tiotropium inhalation powder type A
- Inhaler B, Tiotropium Easyhaler (Experimental): Placebo Tiotropium Easyhaler, type B
  Interventions: Drug: Placebo Tiotropium inhalation powder type B
- Reference product, Spiriva modified HandiHaler (Placebo Comparator): Placebo Spiriva, hard capsule inhaled via modified HandiHaler device
  Interventions: Drug: Placebo Spiriva capsule
- Substudy Test product Placebo Tiotropium Easyhaler (Experimental): The substudy subjects will demonstrate the use of the inhaler.
  Interventions: Device: Substudy Placebo Tiotropium Easyhaler
- Substudy Reference product Placebo Spiriva® HandiHaler (Placebo Comparator): The substudy subjects will demonstrate the use of the inhaler.
  Interventions: Device: Substudy Placebo Spiriva® via HandiHaler

INTERVENTIONS:
Drug: Placebo Tiotropium inhalation powder type A — Placebo inhalation from inhaler A
  Arms: Inhaler A, Tiotropium Easyhaler
Drug: Placebo Spiriva capsule — Placebo inhalation from HandiHaler
  Arms: Reference product, Spiriva modified HandiHaler
Drug: Placebo Tiotropium inhalation powder type B — Placebo inhalation from inhaler B
  Arms: Inhaler B, Tiotropium Easyhaler
Device: Substudy Placebo Tiotropium Easyhaler — Substudy placebo inhalation
  Arms: Substudy Test product Placebo Tiotropium Easyhaler
Device: Substudy Placebo Spiriva® via HandiHaler — Substudy placebo inhalation
  Arms: Substudy Reference product Placebo Spiriva® HandiHaler

SUMMARY:
The study will characterise inspiratory flow parameters across placebo dry powder inhaler Easyhaler (2 inhaler versions) and placebo Spiriva inhalation powder capsule inhaled via HandiHaler in patients with chronic obstructive pulmonary disease (COPD) and in healthy volunteers.

Substudy: Easyhaler® and HandiHaler® Usability study in patients with COPD; to assess patients acceptability, preference, correct use and ability to learn to use Easyhaler and HandiHaler (with capsules) and to compare PIF rate via In-Check Dial meter with the PIF rate via spirometer in the main study.

DETAILED DESCRIPTION:
This is an open, randomised, multicentre, crossover study with Easyhaler and HandiHaler inhalers. The primary objective is to characterise inspiratory flow parameters across placebo dry powder inhaler Easyhaler (2 inhaler versions) and placebo Spiriva inhalation powder capsule inhaled via HandiHaler in patients with chronic obstructive pulmonary disease (COPD) and in healthy volunteers. The secondary objective is to calculate correlation of peak inspiratory flow (PIF) rate with regards to anthropometric and lung function parameters.

Substudy: This is an open, randomised, multicentre, crossover study with Easyhaler and HandiHaler inhalers.There will be 1 study visit per subject, usually this visit is done at the same visit with the main study.

ELIGIBILITY:
Inclusion Criteria for subjects with COPD:

1. Written informed consent (IC) obtained.
2. ≥18 years of age.
3. Documented diagnosis of COPD.

Inclusion Criteria for healthy volunteers:

1. Written informed consent (IC) obtained.
2. ≥18 years of age.
3. FEV1 at least 80% of the predicted value measured at screening.
4. Good general health ascertained by medical history.

Exclusion Criteria for subjects with COPD:

1. Any chronic respiratory disease other than COPD.
2. Acute respiratory infection.
3. Concurrent participation in a clinical drug study.
4. Any medical condition (e.g. contraindications to spirometry) that in the opinion of the investigator could interfere with the interpretation of study results or cause a health risk for the subject if he/she participates in the study. E.g. any concomitant disease in clinically labile state judged by the investigator.
5. Severe milk allergy (lactose contains small amounts of milk proteins).

Exclusion Criteria for healthy volunteers:

1. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic, endocrine, neurological or psychiatric disease within the previous 2 years.
2. Acute respiratory infection.
3. Concurrent participation in a clinical drug study.
4. Any medical condition (e.g. contraindications to spirometry) that in the opinion of the investigator could interfere with the interpretation of study results or cause a health risk for the subject if he/she participates in the study.
5. Severe milk allergy (lactose contains small amounts of milk proteins).

Substudy:

Patients with documented diagnosis of COPD aged 18 year or older participating the main study will be enrolled in this substudy. Written informed consent (IC) will be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
The primary variable will be the PIF rate through the Easyhaler and HandiHaler inhalers. | 1 day
  After practising, 3 inspiratory flow curves will be recorded and the inhalation with the highest PIF rate analysed.

SECONDARY OUTCOMES:
Inspiratory volume through the Easyhaler and HandiHaler inhalers | 1 day
  Highest inspiratory volume recorded and analysed from the same inhalation as the PIF rate.

OTHER OUTCOMES:
Correct use of Easyhaler and HandiHaler tabulated by frequencies and percents based on the inhaler specific questionnaire, assessed by the site staff. | 1 day
  Substudy outcome
Patient's acceptability of inhalers, assessed by the study specific questionnaire | 1 day
  Substudy outcome
Patient's preference of inhalers assessed by study specific questionnaire | 1 day
  Substudy outcome
Patient's ability to learn the use of the inhalers, assessed by the study specific questionnaire. | 1 day
  Substudy outcome
Peak inspiratory flow measurement via In-Check Dial | 1 day
  Substudy outcome

CONTACTS AND LOCATIONS:
Overall Officials: Orion Pharma Clinical Study Director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Lung Clinic, Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kainu A, Vartiainen VA, Mazur W, Hisinger-Molkanen H, Lavorini F, Janson C, Andersson M. Successful Use of Easyhaler(R) Dry Powder Inhaler in Patients with Chronic Obstructive Pulmonary Disease; Analysis of Peak Inspiratory Flow from Three Clinical Trials. Pulm Ther. 2024 Mar;10(1):133-142. doi: 10.1007/s41030-023-00246-8. Epub 2024 Jan 3. PMID 38170393